CLINICAL TRIAL: NCT01773733
Title: All-Russia Non-interventional Program of Reduxine Safety Monitoring for Weight Reduction in Patients With Alimentary Obesity in the Routine Clinical Practice
Brief Title: The PRIMAVERA Study: Reduxine Safety Monitoring in Patients With Alimentary Obesity
Acronym: Primavera
Status: Completed | Type: Observational
Sponsor: Promomed, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: PROMOMED-PRIMAVERA
Record Dates: First submitted 2012-12-20; First posted 2013-01-23 (Estimated); Results first posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2023-04

CONDITIONS: Alimentary Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Obese: Patients 18-65 y.o.with alimentary obesity, BMI (Body Mass Index) ≥ 30 kg/m2)
- Overweight & risk factors: Patients 18-65 y.o., overweight, BMI ≥ 27 kg/m 2 plus T2DM ( type 2 diabetes mellitus) or dyslipidemia

SUMMARY:
The aim of this study is to summarize the data on efficacy and safety of Reduxine administration in the routine clinical practice according to the approved indications.

DETAILED DESCRIPTION:
Secondary objectives:

* to study the structure of the population of patients with the diet induced obesity with body mass index (BMI) 30 kg/m2 or diet induced obesity with BMI ≥27 kg/m2 associated with type 2 diabetes mellitus in respect of comorbidities and concomitant treatment to determine the areas for further investigations.
* to introduce the elements of control of adverse cardiovascular risks into the routine clinical practice: questionnaire concerning enrollment criteria for Reduxine treatment initiation, algorithm of Reduxine administration and treatment efficacy and safety monitoring (assessment schedule).
* to assess the effects of the treatment of overweight and obesity with Reduxine on patients' quality of life parameters.

The Time Frame: the follow up of the study patients will be performed during six month to one year. Exception - premature discontinuation from the study.

The scheduled visits of the patients to the investigational centres are: Week0 (inclusion of the patient), Week 2, 4, 6, 8, 10, 12, 16, 20, 24, 36 and Week 48.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of 18-65 years of age to whom, in the doctor's opinion, the on-label use of Reduxine is indicated.
* Patient's desire and ability to participate in the program and fulfill the doctor's instructions designed to achieve the treatment goal and the program requirements compliance.
* Signed informed consent form for participation in the program.

Exclusion Criteria:

- Patients under age of 18 or older than 65;

Current or the history of:

* coronary artery disease (e.g. angina, myocardial infraction);
* congestive heart failure;
* tachycardia;
* peripheral arterial occlusive disease;
* arrythmia;
* Uncontrolled arterial hypertension >145/90 mm Hg;
* Hypersensitivity to sibutramine or any components of Reduxine®;
* Current use of monoamineoxidase inhibitors (IMAO) or their use within the last 2 weeks;
* Current use of other central acting weight reducing drugs or their use within the last 2 weeks;
* Use on other drugs affecting the central nervous system (e.g. antidepressants, neuroleptics); tryptophan-containing drugs indicated for sleep disturbance;
* Severe eating disorder (anorexia nervosa or bulimia);
* Mental disease;
* Gilles de la Tourette syndrome (generalized tics);
* Body mass index ≤30 kg/m2 or ≤27 kg/m2 in the presence of concomitant diseases (dyslipidemia, diabetes);
* Organic cause of obesity (e.g. hypothyrosis);
* Thyrotoxicosis;
* Sever liver and/or kidney function abnormality;
* Benign prostatic hyperplasia;
* Phaeochromocytoma;
* Narrowangle glaucoma;
* Documented pharmacologic, drug or alcohol addiction;
* Pregnancy and lactation;
* Refusal to sign the informed consent form for participation in the program;
* Participation in a clinical study of any new drug product within 90 days prior to the screening visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women of 18-65 years old, in the random gender and demographical proportion, with the diagnosed overweight (BMI ≥ 27 and < 30) and obesity (BMI ≥ 30).
Sampling Method: Non-Probability Sample
Enrollment: 98774 (Actual)
Dates: Start 2012-11; Primary Completion 2014-07 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivan I Dedov, academician, Study Chair — FEDERAL STATE BUDGETARY INSTITUTION "ENDOCRINOLOGY RESEARCH CENTRE" MINISTRY OF HEALTH OF RUSSIA

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Dedov I.I., Mel'nichenko G.A., Romantsova T.I. The strategy of obesity management: the results of All-Russian observational program "Primavera". Obesity and metabolism. 2016;13(1):36-44. (In Russ.) https://doi.org/10.14341/omet2016136-44
- See also: Obesity and metabolism is peer-reviewed medical journal that publishes articles on the problems of obesity, metabolic disorders, and endocrine diseases — https://www.omet-endojournals.ru/jour/article/view/7988
- Available data/document: published data — https://www.omet-endojournals.ru/jour/article/view/7988 — The observation program allow to implement the principles of active monitoring of the efficacy and safety of the drug in the current clinical practice and to develop a skill of reasonable prescribing. In Primavera program it was shown that the use of Reduxine® (sibutramine+ microcrystalline cellulose) leads to loss of body weight and doesn't lead to serious adverse effect

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 98774 patients signed ICF (Informed Consent Forms), but only 93313 patients started Reduxine treatment, as soon as 5461 patients discontinued prior to the treatment start due to contraindications detected after ICF completion.
Groups:
- Patients With Obesity: Patients 18-65 y.o. with obesity (BMI≥ 30 kg/m2)
- Patients With Overweight Associated With DM2: Patients 18-65 y.o. with DM2 and owerweigt (BMI ≥ 27 kg/m2)
Period: Overall Study
Arm/Group | Patients With Obesity | Patients With Overweight Associated With DM2
Started | 80146 | 13167
3 Months of Treatment | 54841 | 11365
6 Months of Treatment | 33424 | 8007
Completed | 21417 | 4846
Not Completed | 58729 | 8321
Not completed — Adverse Event | 3286 | 540
Not completed — Pregnancy | 28 | 0
Not completed — Other different categories of not compl | 55415 | 7781

BASELINE CHARACTERISTICS:
Groups:
- Patients With Overweight Associated With DM2: Patients 18-65 y.o. with DM2 and overweight (BMI ≥ 27 kg/m2)
- Total: Total of all reporting groups
Arm/Group | Patients With Obesity | Patients With Overweight Associated With DM2 | Total
Number analyzed (Participants) | 80146 | 13167 | 93313
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 80146 | 13167 | 93313
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data for 69810 patients was analyzed. Data for the remaining participants was not analyzed because of the poor quality of Case Report Forms completion.
  Participants
    number analyzed (Participants) | 56643 | 13167 | 69810
    Female | 46617 | 10836 | 57453
    Male | 10026 | 2331 | 12357

OUTCOME MEASURES:

1. Primary Outcome: Body Weight Loss After 3, 6 & 12 Month Treatment
Description: Patients were weighed at each visit, but the statistical data processing was carried out after 3, 6 and 12 months of treatment.
Time Frame: Baseline, after 3, 6 and 12 months of treatment.
Population: Data for 69810 patients was analyzed. Data for the remaining participants was not analyzed because of the poor quality of Case Report Forms completion.
Measure: Mean (Standard Error); unit: kg
Groups:
- Obesity: Patients 18-65 y.o. with alimentary obesity BMI (Body Mass Index) ≥ 30 kg/m2
- Overweight & Risk Factors: Patients 18-65 y.o. overweight, BMI ≥ 27 kg/m2 plus T2DM (type 2 diabetes mellitus) or dyslipidemia
Arm/Group | Obesity | Overweight & Risk Factors
Number analyzed (Participants) | 56643 | 13167
kg
  Body weight loss after 3 month treatment | -9.5 (4.3) | -9.0 (4.19)
  Body weight loss after 6 month treatment: number analyzed (Participants) | 28565 | 12866
  Body weight loss after 6 month treatment | -15.0 (6.2) | -14.4 (5.9)
  Body weight loss after 12 month treatment: number analyzed (Participants) | 21622 | 4641
  Body weight loss after 12 month treatment | -20.0 (8.6) | -19.2 (8.25)

2. Secondary Outcome: Percentage of Participants With Adverse Events
Description: Percentage of participants with all adverse events since the start of the Reduxine treatment to the end of the study
Time Frame: From the 1st day of Reduxine treatment until the end of the treatment
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- Obesity: Patients 18-65 y.o.with alimentary obesity, BMI (Body Mass Index) ≥ 30 kg/m2)
Arm/Group | Obesity | Overweight & Risk Factors
Number analyzed (Participants) | 56643 | 13167
percentage of participants | 4.1 | 4.1
Statistical Analysis 1: Comparison: Obesity vs Overweight & Risk Factors; Test type: Other; p < 0.001, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Obese | Overweight & Risk Factors
All-Cause Mortality (participants affected / at risk) | 0/56643 | 0/13167
Serious Adverse Events (participants affected / at risk) | 0/56643 | 0/13167
Other Adverse Events (participants affected / at risk) | 2322/56643 | 540/13167
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obese (N=56643) | Overweight & Risk Factors (N=13167)
Dry mouth (Nervous system disorders) | 906 (906) | 210 (210)
Headache (General disorders) | 511 (511) | 119 (119) — Headache
Insomnia (Nervous system disorders) | 453 (453) | 105 (105) — Insomnia
Hypertension/increased blood pressure (Cardiac disorders) | 170 (170) | 39 (39) — Hypertension/increased blood pressure
tachycardia (Cardiac disorders) | 114 (114) | 26 (26) — tachycardia
Depression (Nervous system disorders) | 170 (170) | 39 (39) — Depression
Other Adverse Events (General disorders) | 673 (673) | 157 (157) — Other Adverse Events

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No